CLINICAL TRIAL: NCT05518331
Title: Avatrombopag in TPO-RA Refractory Aplastic Anemia Patients Safety and Efficacy Study --Single-arm, Multicenter, Open, Phase Π Clinical Study
Brief Title: The Safety and Efficacy Study of Avatrombopag Switch in TPO-RA Refractory AA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Peking University People's Hospital (Other); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Second Hospital of Shanxi Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Fengkui Zhang, Director of Anemia Treatment Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021008-EC-1
Record Dates: First submitted 2022-06-11; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Refractory Aplastic Anemia
Keywords: Avatrombopag, TPO-RA, refractory aplastic anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — avatrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avatrombopag in RAA (Experimental): After the patients met the above-mentioned inclusion conditions and signed informed consent, they began to be included in this program.
  The main research objectives are to take avatrombopag conversion therapy for at least 3 months, to monitor hematological indicators, biochemical indicators and bone marrow related tests, to determine hematological responses, and to evaluate the safety of the drug.
  In the 6th and 12th months after treatment, comprehensive review of bone marrow and peripheral blood was performed to evaluate the recovery of hematopoiesis, determine the curative effect, evaluate adverse events, and whether there was clonal transformation.
  After the patients completed the main study observation, they were followed up for at least 3 months, that is, from the time the patients were enrolled, for a total of at least 6 months of follow-up.
  Interventions: Drug: avatrombopag

INTERVENTIONS:
Drug: avatrombopag — Avatrombopag, 40-60 mg (body weight < 80 kg, 40 mg per day; body weight > 80 kg, 60 mg per day) orally once daily for at least 3 months and followed up for 3 months to determine hematological response and evaluate the drug security.
  Other Names: CSA

SUMMARY:
This study was a single-arm, multicenter, phase Π clinical study. Patients admitted to the enrollment unit center with a confirmed diagnosis of TDNSAA/VSAA/SAA, treated with IST (p/r-ATG+CSA) in combination with TPO-RA (including eltrombopta or hydtrombopta) for at least 3 months with no hematologic response at 6-month follow-up, and who were not suitable or unwilling to undergo hematopoietic stem cell transplantation (HSCT), were to another novel TPO-RA avatrombopta, 40-60 mg (weight <80 kg), in addition to maintaining the original immunosuppressive therapy ( CSA or equivalent immune potency drugs), switch to another new TPO-RA avatropa 40-60 mg (40 mg daily for weight <80 kg; 60 mg daily for weight >80 kg) orally once daily for at least 3 months and follow up for 3 months to determine the hematologic response and to assess the safety of the drug

DETAILED DESCRIPTION:
This study was a single-arm, multicenter, phase Π clinical study. Patients admitted to the enrollment unit center with a confirmed diagnosis of TDNSAA/VSAA/SAA, treated with IST (p/r-ATG+CSA) in combination with TPO-RA (including eltrombopta or hydtrombopta) for at least 3 months with no hematologic response at 6-month follow-up, and who were not suitable or unwilling to undergo hematopoietic stem cell transplantation (HSCT), were to another novel TPO-RA avatrombopta, 40-60 mg (weight <80 kg), in addition to maintaining the original immunosuppressive therapy ( CSA or equivalent immune potency drugs), switch to another new TPO-RA avatropa 40-60 mg (40 mg daily for weight <80 kg; 60 mg daily for weight >80 kg) orally once daily for at least 3 months and follow up for 3 months to determine the hematologic response and to assess the safety of the drug.Selection of study population Severe aplastic anemia patients with poor efficacy of IST combined with TPO-RA Patients should be judged for inclusion and exclusion criteria. Number of subjects: 35 effective cases, 39 patients should be included according to the dropout rate of 10%.

ELIGIBILITY:
Inclusion Criteria: Subjects eligible for inclusion in this study must meet all of the following criteria:

1. Patients with confirmed TDNSAA/SAA/VSAA aplastic anemia who received standard IST therapy for at least 6 months, combined with Haitrombopag (15mg/d) or Eltrombopag (>50mg/d) for at least 3 Patients who have not obtained a hematological response (NR) for months and are not suitable or unwilling to undergo HSCT
2. Age > 14 years old, male or female.
3. Subjects must complete all screening assessments listed in the trial protocol.
4. ECOG score ≤ 2 points.
5. Before the start of the research procedure, the patient or guardian should fully understand the research procedure and purpose and sign the informed consent form. If the patient's signature is not conducive to the treatment of the disease, the patient's immediate family should sign the informed consent form.

Exclusion Criteria: Subjects meeting any of the following criteria were excluded from this study:

1. Patients with severe infectious diseases (uncured tuberculosis, pulmonary aspergillosis, various bacterial and viral infections) and active bleeding that cannot be controlled after standard treatment.
2. Patients with AIDS, active viral hepatitis B, and hepatitis C RNA nucleic acid test positive.
3. Those who are pregnant or breastfeeding, have fertility but are unwilling to take effective contraceptive measures.
4. Congenital hematopoietic failure diseases (such as Fanconi anemia).
5. Patients with cytogenetic clonal changes (excluding germline mutations and acquired chromosome clones of +8, 20q- and -y).
6. Combined with malignant tumor within 3 years.
7. Combined with other systemic diseases that cannot be controlled.
8. Significant abnormalities in cardiopulmonary function.
9. Abnormal liver and kidney function: creatinine level > 1.5 times the upper limit of normal, transaminase and bilirubin level > 2 times the upper limit of normal, and those who cannot be enrolled in the group as judged by the clinician.
10. Those who are considered unsuitable for enrollment by the investigator.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The rate of HR in patients after switching to avatrombopag. | 3 months
  Percentage of the total number of patients receiving treatment who received APAG
Incidence of Treatment-Emergent Adverse Events as assessed by information on Common Toxicity Criteria (CTC) AE grading | 3 months
  Incidence of Treatment-Emergent AE by CTCAE
Percentage of patients with transformation | 3 months
  Rate of patients with transformation to PNH or MDS,AML, or other disease

SECONDARY OUTCOMES:
The rate of HR in patients after switching to avatrombopag. | 6months
  Percentage of the total number of patients receiving treatment who received APAG
ncidence of Treatment-Emergent Adverse Events as assessed by information on Common Toxicity Criteria (CTC) AE grading | 6months
  Incidence of Treatment-Emergent AE by CTCAE
Percentage of patients with transformation | 6months
  Rate of patients with transformation to PNH or MDS,AML, or other disease
The rate of HR in patients after switching to avatrombopag. | 12months
  Percentage of the total number of patients receiving treatment who received APAG
ncidence of Treatment-Emergent Adverse Events as assessed by information on Common Toxicity Criteria (CTC) AE grading | 12months
  Incidence of Treatment-Emergent AE by CTCAE
Percentage of patients with transformation | 12months
  Rate of patients with transformation to PNH or MDS,AML, or other disease

CONTACTS AND LOCATIONS:
Overall Officials: Liping Jing, Doctor, Study Director — Anemia Treatment Center
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We can share the plan after completing the experiment
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Follow-up and publication of the paper are planned for December 2025
Access Criteria: After the paper is written and published

REFERENCES:
- [Result] Killick SB, Bown N, Cavenagh J, Dokal I, Foukaneli T, Hill A, Hillmen P, Ireland R, Kulasekararaj A, Mufti G, Snowden JA, Samarasinghe S, Wood A, Marsh JC; British Society for Standards in Haematology. Guidelines for the diagnosis and management of adult aplastic anaemia. Br J Haematol. 2016 Jan;172(2):187-207. doi: 10.1111/bjh.13853. Epub 2015 Nov 16. No abstract available. PMID 26568159
- [Result] Scheinberg P. Activity of eltrombopag in severe aplastic anemia. Hematology Am Soc Hematol Educ Program. 2018 Nov 30;2018(1):450-456. doi: 10.1182/asheducation-2018.1.450. PMID 30504345
- [Result] Townsley DM, Scheinberg P, Winkler T, Desmond R, Dumitriu B, Rios O, Weinstein B, Valdez J, Lotter J, Feng X, Desierto M, Leuva H, Bevans M, Wu C, Larochelle A, Calvo KR, Dunbar CE, Young NS. Eltrombopag Added to Standard Immunosuppression for Aplastic Anemia. N Engl J Med. 2017 Apr 20;376(16):1540-1550. doi: 10.1056/NEJMoa1613878. PMID 28423296
- [Result] Olnes MJ, Scheinberg P, Calvo KR, Desmond R, Tang Y, Dumitriu B, Parikh AR, Soto S, Biancotto A, Feng X, Lozier J, Wu CO, Young NS, Dunbar CE. Eltrombopag and improved hematopoiesis in refractory aplastic anemia. N Engl J Med. 2012 Jul 5;367(1):11-9. doi: 10.1056/NEJMoa1200931. PMID 22762314
- [Result] Peng G, He G, Chang H, Gao S, Liu X, Chen T, Li P, Han B, Miao M, Ge Z, Ge X, Li F, Li Y, Wang S, Wang Y, Shen Y, Zhang T, Zou J, Zhang F. A multicenter phase II study on the efficacy and safety of hetrombopag in patients with severe aplastic anemia refractory to immunosuppressive therapy. Ther Adv Hematol. 2022 Mar 30;13:20406207221085197. doi: 10.1177/20406207221085197. eCollection 2022. PMID 35371427
- [Result] Ise M, Iizuka H, Kamoda Y, Hirao M, Kida M, Usuki K. Romiplostim is effective for eltrombopag-refractory aplastic anemia: results of a retrospective study. Int J Hematol. 2020 Dec;112(6):787-794. doi: 10.1007/s12185-020-02971-1. Epub 2020 Sep 2. PMID 32876852